CLINICAL TRIAL: NCT02687711
Title: A 12-Month Noninterventional, Postmarketing, Multicenter Study to Evaluate the Effectiveness of Briviact® (Brivaracetam) as Adjunctive Therapy in Patients With Epilepsy With Partial-onset Seizures in Daily Clinical Practice
Brief Title: Study to Look at How Effective Briviact is as add-on Treatment for Patients With Epilepsy With Partial Onset Seizures
Acronym: BASE
Status: Completed | Type: Observational
Sponsor: UCB Biopharma S.P.R.L. (Industry)
Collaborators: Pharm Research Associates Ltd. UK (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Other Study IDs: EP0077
Record Dates: First submitted 2016-02-12; First posted 2016-02-22 (Estimated); Results first posted 2021-08-04 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-07

CONDITIONS: Epilepsy With POS With or Without Secondary Generalization
Keywords: Non-interventional (NIS); Epilepsy; Partial Onset Seizures (POS); add-on therapy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Study is the first study after commercialization of brivaracetam. It is designed to collect real world information on the effectiveness of brivaracetam in patients with Partial Onset Seizure epislepsy who are treated in standard clinical practice.

DETAILED DESCRIPTION:
EP0077 is a 12 months, multicenter, noninterventional study (NIS) conducted at specialized sites in approximately 10 European countries. Patients will be treated according to usual medical diagnostic procedures and therapy; commercially available brivaracetam will be prescribed according to normal clinical practice and the current Summary of Product Characteristics (SmPC) in Europe for brivaracetam (BRV). The prescription of BRV is clearly separated from the decision to include the patient in the study. No additional diagnostic or monitoring procedures are applied to the patients.

The primary objective of this study is to determine BRV retention over a 12 month period as a measure of effectiveness in a real world setting. The secondary objective of this study is to assess seizure control with BRV treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patient has never been treated with brivaracetam (BRV) prior to enrollment in this Non-Interventional Study (NIS)
* The decision by the treating physician to prescribe BRV is made independently of the participation in the NIS
* Patient is a male or female ≥16 years of age
* Patient has a clinical diagnosis of epilepsy with partial-onset seizures POS with or without secondary generalization
* Patient uses an epilepsy/seizure diary.

Exclusion Criteria:

No specific exclusion criteria

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients (male or female ≥16 years of age) with a clinical diagnosis of epilepsy with Partial Onset Seizures with or without secondary generalization. The patients have never been treated with brivaracetam and the decision by the treating physician (neurologists) to prescribe brivaracetam is made independently of the participation in the study and prior to enrollment.
  Patient meets the criteria for treatment with brivaracetam as adjunctive therapy according to the current SmPC in Europe. Patient is using a seizure diary as part of their standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 544 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — +1 844 599 2273 (UCB)
Locations (44):
- Denmark (3):
  - Ep0077 4504, Aarhus
  - Ep0077 4501, Glostrup Municipality
  - Ep0077 4503, Odense
- Germany (8):
  - Ep0077 4906, Berlin
  - Ep0077 4910, Bonn
  - Ep0077 4909, Freiburg im Breisgau
  - Ep0077 4913, Hamburg
  - Ep0077 4901, Kork
  - Ep0077 4912, Radeberg
  - Ep0077 4904, Ravensburg
  - Ep0077 4905, Tübingen
- Hungary (6):
  - Ep0077 3605, Budapest
  - Ep0077 3608, Kecskemét
  - Ep0077 3607, Mosdós
  - Ep0077 3602, Nyíregyháza
  - Ep0077 3601, Pécs
  - Ep0077 3606, Szeged
- Ireland (3):
  - Ep0077 3503, Cork
  - Ep0077 3501, Dublin
  - Ep0077 3505, Dublin
- Italy (4):
  - Ep0077 3912, Florence
  - Ep0077 3901, Milan
  - Ep0077 3904, Milan
  - Ep0077 3902, Verona
- Netherlands (2):
  - Ep0077 3101, Heeze
  - Ep0077 3102, Maastricht
- Ep0077 4701, Fredrikstad, Norway
- Spain (4):
  - Ep0077 3402, A Coruña
  - Ep0077 3416, Badajoz
  - Ep0077 3412, Córdoba
  - Ep0077 3410, Murcia
- United Kingdom (13):
  - Ep0077 4408, Birmingham
  - Ep0077 4414, Cardiff
  - Ep0077 4406, Dundee
  - Ep0077 4401, Glasgow
  - Ep0077 4417, Inverness
  - Ep0077 4404, Leeds
  - Ep0077 4409, London
  - Ep0077 4411, London
  - Ep0077 4403, Salford
  - Ep0077 4407, Sheffield
  - Ep0077 4412, Stoke-on-Trent
  - Ep0077 4416, Swansea
  - Ep0077 4402, Truro

IPD SHARING:
Plan to Share IPD: No
Data from non-interventional studies is outside of UCB's data sharing policy and is unavailable for sharing.

REFERENCES:
- See also: Product Information — http://www.briviact.com/briviact-PI.pdf?v=1479491757
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll participants in February 2016 and concluded in July 2020.
Pre-assignment Details: Participant Flow refers to the Safety Set.
Groups:
- Brivaracetam (BRV): Participants were treated with commercially available BRV as prescribed by treating physicians, in accordance with current clinical practice and in accordance with the approved European Summary of Product Characteristics (SmPC).
Period: Overall Study
Arm/Group | Brivaracetam (BRV)
Started | 544
Completed | 332
Not Completed | 212
Not completed — Adverse Event | 89
Not completed — Lack of Efficacy | 70
Not completed — Lost to Follow-up | 20
Not completed — Consent withdrawn | 15
Not completed — Participant moved to another country and continued treatment for epilepsy in that country | 1
Not completed — Too expensive | 4
Not completed — Participant moved abroad | 1
Not completed — Progression of other medical condition (dementia, pneumonia) | 1
Not completed — Perceived increase in seizures but diary records show no increase compared to pre-study | 1
Not completed — Disliked taste | 1
Not completed — Low mood | 1
Not completed — Side effects | 1
Not completed — Change of Hospital | 1
Not completed — Liver Encephalopathy | 1
Not completed — Participant experience side effects, fatigue. Most likely not related to investigational product | 1
Not completed — Withdrawn due to intake interruption | 1
Not completed — Stopped in preparation for epilepsy surgery | 1
Not completed — Diagnosis epilepsy revised to psychogenic seizures | 1
Not completed — Participant was not able to come in our clinic because participant could not find a car driver | 1

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Safety Set which consisted of all participants which were included in the All Subjects Documented Set for whom it could not be excluded that they received treatment with BRV at least once in the study.
Arm/Group | Brivaracetam (BRV)
Number analyzed (Participants) | 544
Age, Categorical [Count of Participants; unit: Participants] — Baseline Characteristics refer to the Safety Set which consisted of all participants which were included in the All Subjects Documented Set for whom it could not be excluded that they received treatment with BRV at least once in the study.
  Participants
    <=18 years | 8
    Between 18 and 65 years | 492
    >=65 years | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.6 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 287
  Male | 257
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Remaining in the Study and on BRV Treatment at Month 12
Description: Participants who remained in the study and were on BRV treatment for at least 1 year (>=330 days) after their start of BRV were classed as having 12 months of treatment retention.
Time Frame: Month 12 (end of Observation Period)
Population: The Full Analysis Set (FAS) was defined as all participants in the Safety Set (SS) who did not receive BRV before entering this non interventional study (NIS).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Brivaracetam (FAS): Participants were treated with commercially available BRV as prescribed by treating physicians, in accordance with current clinical practice and in accordance with the approved European Summary of Product Characteristics (SmPC). Participants formed the Full Analysis Set (FAS).
Arm/Group | Brivaracetam (FAS)
Number analyzed (Participants) | 541
percentage of participants | 57.7 [53.4 to 61.9]

2. Secondary Outcome: Percentage of Participants Remaining in the Study and on BRV Treatment at Month 3
Description: Participants who remained in the study and were on BRV treatment for at least 3 months (>=90 days) after first BRV administration were classed as having 3 months of treatment retention.
Time Frame: Month 3
Population: FAS was defined as all participants in the Safety Set (SS) who did not receive BRV before entering this NIS.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Brivaracetam (FAS)
Number analyzed (Participants) | 541
percentage of participants | 82.4 [79.0 to 85.6]

3. Secondary Outcome: Percentage of Participants Remaining in the Study and on BRV Treatment at Month 6
Description: Participants who remained in the study and were on BRV treatment for at least 6 months (>=180 days) after first BRV administration were classed as having 6 months of treatment retention.
Time Frame: Month 6
Population: FAS was defined as all participants in the Safety Set (SS) who did not receive BRV before entering this NIS.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Brivaracetam (FAS)
Number analyzed (Participants) | 541
percentage of participants | 70.6 [66.6 to 74.4]

4. Secondary Outcome: Absolute Change in Partial-onset Seizure (POS) Frequency From Baseline to Month 3
Description: Absolute change in POS frequency was defined as: 28-day Baseline - 28-day post-Baseline seizure frequency.
Time Frame: From Baseline (Day 1) to Month 3
Population: FAS was defined as all participants in the Safety Set (SS) who did not receive BRV before entering this NIS. Here number of participants were included who were evaluable for the assessment.
Measure: Mean (Standard Deviation); unit: seizures per 28 days
Arm/Group | Brivaracetam (FAS)
Number analyzed (Participants) | 398
seizures per 28 days | 4.54 (24.34)

5. Secondary Outcome: Absolute Change in Partial-onset Seizure (POS) Frequency From Baseline to Month 6
Description: Absolute change in POS frequency was defined as: 28-day Baseline - 28-day post-Baseline seizure frequency.
Time Frame: From Baseline (Day 1) to Month 6
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: seizures per 28 days
Arm/Group | Brivaracetam (FAS)
Number analyzed (Participants) | 343
seizures per 28 days | 3.29 (16.92)

6. Secondary Outcome: Absolute Change in Partial-onset Seizure (POS) Frequency From Baseline to Month 12
Description: Absolute change in POS frequency was defined as: 28-day Baseline - 28-day post-Baseline seizure frequency.
Time Frame: From Baseline (Day 1) to Month 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: seizures per 28 days
Arm/Group | Brivaracetam (FAS)
Number analyzed (Participants) | 259
seizures per 28 days | 3.75 (16.05)

7. Secondary Outcome: Absolute Change in Partial-onset Seizure (POS) Frequency From Baseline to End of Observation Period
Description: Absolute change in POS frequency was defined as: 28-day Baseline - 28-day post-Baseline seizure frequency.
Time Frame: From Baseline (Day 1) to end of Observation Period (up to Month 12/withdrawal)
Population: FAS was defined as all participants in the Safety Set (SS) who did not receive BRV before entering this NIS. Here number of participants were included who were evaluable for the assessment and were classified as study completers or who withdrew early.
Measure: Mean (Standard Deviation); unit: seizures per 28 days
Arm/Group | Brivaracetam (FAS)
Number analyzed (Participants) | 373
seizures per 28 days | 1.69 (26.59)

8. Secondary Outcome: Percent Change in Partial-onset Seizure (POS) Frequency From Baseline to Month 3
Description: Percent change in POS frequency was defined as: ((28-day Baseline - 28-day post-Baseline seizure frequency)/28-day Baseline) x 100. A positive value indicates a reduction.
Time Frame: From Baseline (Day 1) to Month 3
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Brivaracetam (FAS)
Number analyzed (Participants) | 362
percent change | -5.39 (215.31)

9. Secondary Outcome: Percent Change in Partial-onset Seizure (POS) Frequency From Baseline to Month 6
Description: as for outcome 8
Time Frame: From Baseline (Day 1) to Month 6
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Brivaracetam (FAS)
Number analyzed (Participants) | 308
percent change | -10.64 (369.03)

10. Secondary Outcome: Percent Change in Partial-onset Seizure (POS) Frequency From Baseline to Month 12
Description: as for outcome 8
Time Frame: From Baseline (Day 1) to Month 12
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Brivaracetam (FAS)
Number analyzed (Participants) | 230
percent change | 7.05 (351.75)

11. Secondary Outcome: Percent Change in Partial-onset Seizure (POS) Frequency From Baseline to End of Observation Period
Description: as for outcome 8
Time Frame: From Baseline (Day 1) to end of Observation Period (up to Month 12/withdrawal)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Brivaracetam (FAS)
Number analyzed (Participants) | 339
percent change | -9.54 (308.89)

12. Secondary Outcome: Number of Responders Based on Percent Reduction (>=50%) in Partial-onset Seizure (POS) Frequency at Month 3
Description: Response was defined as a (greater than or equal to [>=] 50%) reduction from Baseline in seizure frequency.
Time Frame: Baseline (Day 1) to Month 3
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Brivaracetam (FAS)
Number analyzed (Participants) | 362
Participants | 170

13. Secondary Outcome: Percent of Responders Based on Percent Reduction (>=50%) in Partial-onset Seizure (POS) Frequency at Month 3
Description: Response was defined as a >=50% reduction from Baseline in seizure frequency.
Time Frame: Baseline (Day 1) to Month 3
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Brivaracetam (FAS)
Number analyzed (Participants) | 362
percentage of participants | 47.0

14. Secondary Outcome: Number of Responders Based on Percent Reduction (>=50%) in Partial-onset Seizure (POS) Frequency at Month 6
Description: Response was defined as a >=50% reduction from Baseline in seizure frequency.
Time Frame: Baseline (Day 1) to Month 6
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Brivaracetam (FAS)
Number analyzed (Participants) | 308
Participants | 146

15. Secondary Outcome: Percent of Responders Based on Percent Reduction (>=50%) in Partial-onset Seizure (POS) Frequency at Month 6
Description: Response was defined as a >=50% reduction from Baseline in seizure frequency.
Time Frame: Baseline (Day 1) to Month 6
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Brivaracetam (FAS)
Number analyzed (Participants) | 308
percentage of participants | 47.4

16. Secondary Outcome: Number of Responders Based on Percent Reduction (>=50%) in Partial-onset Seizure (POS) Frequency at Month 12
Description: Response was defined as a >=50% reduction from Baseline in seizure frequency.
Time Frame: Baseline (Day 1) to Month 12
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Brivaracetam (FAS)
Number analyzed (Participants) | 230
Participants | 139

17. Secondary Outcome: Percent of Responders Based on Percent Reduction (>=50%) in Partial-onset Seizure (POS) Frequency at Month 12
Description: Response was defined as a >=50% reduction from Baseline in seizure frequency.
Time Frame: Baseline (Day 1) to Month 12
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Brivaracetam (FAS)
Number analyzed (Participants) | 230
percentage of participants | 60.4

18. Secondary Outcome: Number of Responders Based on Percent Reduction (>=50%) in Partial-onset Seizure (POS) Frequency at End of Observation Period
Description: Response was defined as a >=50% reduction from Baseline in seizure frequency.
Time Frame: Baseline (Day 1) to end of Observation Period (up to Month 12/withdrawal)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Brivaracetam (FAS)
Number analyzed (Participants) | 339
Participants | 175

19. Secondary Outcome: Percent of Responders Based on Percent Reduction (>=50%) in Partial-onset Seizure (POS) Frequency at End of Observation Period
Description: Response was defined as a >=50% reduction from Baseline in seizure frequency.
Time Frame: Baseline (Day 1) to end of Observation Period (up to Month 12/withdrawal)
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | Brivaracetam (FAS)
Number analyzed (Participants) | 339
percentage of participants | 51.6

20. Secondary Outcome: Number of Seizure Free Participants (When Discontinuations Were Counted as Seizure Freedom=no) at Month 3
Description: Seizure freedom (Yes) was defined as having no seizures recorded in the study on or before the visit date, having not discontinued prior to the visit and having available seizure data at the visit. Participants with seizures before the visit date or participants who discontinued BRV or terminated the study prior to the target visit date (Visit 2 [Month 3] = Day 90) were counted as No.
Time Frame: Month 3
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Brivaracetam (FAS)
Number analyzed (Participants) | 497
Participants | 81

21. Secondary Outcome: Percent of Seizure Free Participants (When Discontinuations Were Counted as Seizure Freedom=no) at Month 3
Description: as for outcome 20
Time Frame: Month 3
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Brivaracetam (FAS)
Number analyzed (Participants) | 497
percentage of participants | 16.3

22. Secondary Outcome: Number of Seizure Free Participants (When Discontinuations Were Counted as Seizure Freedom=Missing) at Month 3
Description: Seizure freedom (Yes) was defined as having no seizures recorded in the study on or before the visit date, having not discontinued prior to the visit and having available seizure data at the visit. Participants with seizures before the visit date were counted as a No. Participants who discontinued BRV or terminated the study prior to the target visit date without any seizures recorded up to discontinuation or termination were excluded from the analysis.
Time Frame: Month 3
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Brivaracetam (FAS)
Number analyzed (Participants) | 454
Participants | 81

23. Secondary Outcome: Percent of Seizure Free Participants (When Discontinuations Were Counted as Seizure Freedom=Missing) at Month 3
Description: as for outcome 22
Time Frame: Month 3
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Brivaracetam (FAS)
Number analyzed (Participants) | 454
percentage of participants | 17.8

24. Secondary Outcome: Number of Seizure Free Participants (When Discontinuations Were Counted as Seizure Freedom=no) at Month 6
Description: Seizure freedom (Yes) was defined as having no seizures recorded in the study on or before the visit date, having not discontinued prior to the visit and having available seizure data at the visit. Participants with seizures before the visit date or participants who discontinued BRV or terminated the study prior to the target visit date (Visit 3 [Month 6] = Day 180) were counted as No.
Time Frame: Month 6
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Brivaracetam (FAS)
Number analyzed (Participants) | 510
Participants | 54

25. Secondary Outcome: Percent of Seizure Free Participants (When Discontinuations Were Counted as Seizure Freedom=no) at Month 6
Description: as for outcome 24
Time Frame: Month 6
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Brivaracetam (FAS)
Number analyzed (Participants) | 510
percentage of participants | 10.6

26. Secondary Outcome: Number of Seizure Free Participants (When Discontinuations Were Counted as Seizure Freedom=Missing) at Month 6
Description: as for outcome 22
Time Frame: Month 6
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Brivaracetam (FAS)
Number analyzed (Participants) | 456
Participants | 54

27. Secondary Outcome: Percent of Seizure Free Participants (When Discontinuations Were Counted as Seizure Freedom=Missing) at Month 6
Description: as for outcome 22
Time Frame: Month 6
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Brivaracetam (FAS)
Number analyzed (Participants) | 456
percentage of participants | 11.8

28. Secondary Outcome: Number of Seizure Free Participants (When Discontinuations Were Counted as Seizure Freedom=no) at Month 12
Description: Seizure freedom (Yes) was defined as having no seizures recorded in the study on or before the visit date, having not discontinued prior to the visit and having available seizure data at the visit. Participants with seizures before the visit date or participants who discontinued BRV or terminated the study prior to the target visit date (Visit 4 [Month 12] = Day 330) were counted as No.
Time Frame: Month 12
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Brivaracetam (FAS)
Number analyzed (Participants) | 269
Participants | 37

29. Secondary Outcome: Percent of Seizure Free Participants (When Discontinuations Were Counted as Seizure Freedom=no) at Month 12
Description: as for outcome 28
Time Frame: Month 12
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Brivaracetam (FAS)
Number analyzed (Participants) | 269
percentage of participants | 13.8

30. Secondary Outcome: Number of Seizure Free Participants (When Discontinuations Were Counted as Seizure Freedom=Missing) at Month 12
Description: as for outcome 22
Time Frame: Month 12
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Brivaracetam (FAS)
Number analyzed (Participants) | 269
Participants | 37

31. Secondary Outcome: Percent of Seizure Free Participants (When Discontinuations Were Counted as Seizure Freedom=Missing) at Month 12
Description: as for outcome 22
Time Frame: Month 12
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Brivaracetam (FAS)
Number analyzed (Participants) | 269
percentage of participants | 13.8

32. Secondary Outcome: Time to First Seizure After First Dose of Brivaracetam
Description: Time to first seizure was calculated as: Date of first seizure - date of first BRV administration + 1.
Time Frame: Month 12
Population: FAS was defined as all participants in the Safety Set (SS) who did not receive BRV before entering this NIS.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Brivaracetam (FAS)
Number analyzed (Participants) | 541
days | 15 [11 to 20]

33. Secondary Outcome: Number of Seizure Free Participants at End of Observation Period
Description: Seizure freedom (Yes) was defined as having no seizures recorded in the study on or before the visit date, having not discontinued prior to the visit and having available seizure data at the visit. End of Observation Period (up to Month 12), includes participants who are completers or withdrew early.
Time Frame: End of Observation Period (up to Month 12/withdrawal)
Population: FAS was defined as all participants in the Safety Set (SS) who did not receive BRV before entering this NIS.
Measure: Count of Participants; unit: Participants
Arm/Group | Brivaracetam (FAS)
Number analyzed (Participants) | 541
Participants | NA — There was no opportunity for the participant to withdraw from the study at the 12-month time point, as they were classified as completers at that stage. Therefore, by definition End of Observation Period (up to Month 12, which includes participants as withdrawn or completers) was identical to Month 12 (including completers alone) results. Hence, the analysis were not performed for this outcome measure.

34. Secondary Outcome: Percent of Seizure Free Participants at End of Observation Period
Description: as for outcome 33
Time Frame: End of Observation Period (up to Month 12/withdrawal)
Population: FAS was defined as all participants in the Safety Set (SS) who did not receive BRV before entering this NIS.
Measure: Number; unit: percentage of participants
Arm/Group | Brivaracetam (FAS)
Number analyzed (Participants) | 541
percentage of participants | NA — There was no opportunity for the participant to withdraw from the study at the 12-month time point, as they were classified as completers at that stage. Therefore, by definition End of Observation Period (up to Month 12, which includes participants as withdrawn or completers) was identical to Month 12 (including completers alone) results. Hence, the analysis were not performed for this outcome measure.

ADVERSE EVENTS:
Time Frame: From Baseline up to Month 12
Description: Treatment-emergent adverse events (TEAEs) were defined as an adverse event (AE) occurring on or after the date of first BRV administration.
Groups:
- Brivaracetam (SS): Participants were treated with commercially available BRV as prescribed by treating physicians, in accordance with current clinical practice and in accordance with the approved European Summary of Product Characteristics (SmPC). Participants formed the Safety Set (SS).
Arm/Group | Brivaracetam (SS)
All-Cause Mortality (participants affected / at risk) | 2/544
Serious Adverse Events (participants affected / at risk) | 80/544
Other Adverse Events (participants affected / at risk) | 62/544
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brivaracetam (SS) (N=544)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Cleft lip (Congenital, familial and genetic disorders) | 1 (1)
Cleft palate (Congenital, familial and genetic disorders) | 1 (1)
Diplopia (Eye disorders) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Oesophageal rupture (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Death (General disorders) | 2 (2)
Malaise (General disorders) | 2 (2)
Drug intolerance (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2)
Actinomycosis (Infections and infestations) | 1 (1)
Empyema (Infections and infestations) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 1 (1)
Streptococcal sepsis (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Burns third degree (Injury, poisoning and procedural complications) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1)
Soft tissue injury (Injury, poisoning and procedural complications) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1)
Clinical global impression scale (Investigations) | 1 (1)
Electroencephalogram (Investigations) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Seizure (Nervous system disorders) | 30 (31)
Generalised tonic-clonic seizure (Nervous system disorders) | 8 (8)
Partial seizures (Nervous system disorders) | 4 (4)
Epilepsy (Nervous system disorders) | 3 (3)
Seizure cluster (Nervous system disorders) | 3 (3)
Focal dyscognitive seizures (Nervous system disorders) | 2 (2)
Petit mal epilepsy (Nervous system disorders) | 2 (2)
Status epilepticus (Nervous system disorders) | 2 (2)
Change in seizure presentation (Nervous system disorders) | 1 (1)
Cognitive disorder (Nervous system disorders) | 1 (1)
Dementia Alzheimer's type (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 1 (1)
Postictal state (Nervous system disorders) | 1 (1)
Tonic convulsion (Nervous system disorders) | 1 (1)
Gestational diabetes (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 9 (9)
Aggression (Psychiatric disorders) | 6 (6)
Affective disorder (Psychiatric disorders) | 2 (2)
Agitation (Psychiatric disorders) | 2 (2)
Mood altered (Psychiatric disorders) | 2 (2)
Anger (Psychiatric disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Behaviour disorder (Psychiatric disorders) | 1 (1)
Depressed mood (Psychiatric disorders) | 1 (1)
Drug abuse (Psychiatric disorders) | 1 (1)
Mood swings (Psychiatric disorders) | 1 (1)
Paranoia (Psychiatric disorders) | 1 (1)
Personality change (Psychiatric disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Abortion induced (Surgical and medical procedures) | 1 (1)
Epilepsy surgery (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brivaracetam (SS) (N=544)
Drug ineffective (General disorders) | 62 (63)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-10-25): https://cdn.clinicaltrials.gov/large-docs/11/NCT02687711/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-09): https://cdn.clinicaltrials.gov/large-docs/11/NCT02687711/SAP_001.pdf